CLINICAL TRIAL: NCT07080515
Title: Developing an Approach to Implementing Breast Cancer Screening Using Clinical Breast Exam in the Primary Health Centers of Abuja, Nigeria
Brief Title: Developing Screening Clinical Breast Examination Implementation Strategies in Nigeria
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: 2000040678; K08CA279913 (NIH)
Record Dates: First submitted 2025-06-30; First posted 2025-07-23 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Detection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adopters: Individuals responsible for deciding to institute screening CBE in Abuja's primary care clinics (e.g., policymakers, clinic administrators, nurse managers)
- Implementers: Individuals responsible for actually performing the screening CBE in Abuja's primary care clinics (e.g., nurses, doctors, fieldworkers, clerical workers)
- Recipients: Individuals eligible for a screening CBE (e.g., women over the age of 40 years from the community surrounding study clinics)

SUMMARY:
The goal of this observational study is to engage with multilevel stakeholders to collaboratively and to systematically develop a suite of strategies for implementing breast cancer screening using clinical breast examination (CBE) in the primary health centers of Abuja, Nigeria.

The main questions it aims to answer are: What barriers and facilitators exist to conducting screening CBE in Abuja's primary care setting and what implementation strategies would support CBE in primary care clinics?

Participants will:

* Allow observation of study clinic workflows
* Participate in interviews and focus group discussions regarding screening CBE implementation

ELIGIBILITY:
In order to be eligible for inclusion in the focus group discussions held with screening CBE "adopters" and "implementers," an individual must meet all of the following criteria:

1. Be an employee or volunteer working at a participating PHC OR Be an employee or volunteer working at Nigeria's Ministry of Health OR Be an employee or volunteer working with a non-governmental organization that performs breast cancer related activities within the catchment area of a participating PHC
2. Be willing to commit to keeping the content of focus group discussions confidential

In order to be eligible for inclusion in the focus group discussions held with screening CBE "recipients," an individual must meet all of the following criteria:

1. Be female
2. Be between the ages of 40 and 65 years
3. Be living within the catchment area of a participating PHC
4. Be willing to commit to keeping the content of focus group discussions confidential

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Focus group participants will consist of three categories: screening CBE "adopter" (e.g., clinic administrators/managers, department of health officials, etc), "implementers" (e.g., nurses, physicians, community health workers), and "recipients" (e.g., women from the community eligible for CBE screening and community breast cancer survivors).
  All participants will be drawn from the two study clinics in Abuja, Nigeria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Domain Characteristics | 1 year
  Characteristics of routine clinical breast examination itself that are potential barriers and facilitators to screening implementation, emerging from thematic analysis of qualitative data organized according to the Consolidated Framework for Implementation Research.
Inner Setting Domain Characteristics | 1 year
  Characteristics of the primary care clinics that are potential barriers and facilitators to screening implementation, emerging from thematic analysis of qualitative data organized according to the Consolidated Framework for Implementation Research.
Outer Setting Domain Characteristics | 1 year
  Characteristics of both the community surrounding the clinics and the district-wide health system that are potential barriers and facilitators to screening implementation, , emerging from thematic analysis of qualitative data organized according to the Consolidated Framework for Implementation Research.
Individuals Domain Characteristics | 1 year
  Characteristics of individuals involved in screening that are potential barriers and facilitators to screening implementation, emerging from thematic analysis of qualitative data organized according to the Consolidated Framework for Implementation Research.
Implementation Domain Characteristics | 1 year
  Characteristics of activities and strategies used to implement screening that are potential barriers and facilitators to screening implementation, emerging from thematic analysis of qualitative data organized according to the Consolidated Framework for Implementation Research.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O'Neil, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Institute of Human Virology, Nigeria, Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: No
In order to comply with local legal requirements, individual participant data will not be available to other researchers.